CLINICAL TRIAL: NCT05414786
Title: A Phase 1 Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) in HIV-1 Uninfected Adults in Good General Health
Brief Title: A Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: AURUM Tembisa Clinical Research (Unknown); Center for Family Health Research (Unknown); ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IAVI G003
Record Dates: First submitted 2022-05-26; First posted 2022-06-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection
Keywords: eOD-GT8 60mer mRNA Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): * 2 doses eOD-GT8 60mer mRNA Vaccine (100µg), 2 vaccinations, 8 weeks apart
  * No control group. There is no blinding and no randomization in this open label study
  Interventions: Biological: eOD-GT8 60mer mRNA Vaccine (100µg)

INTERVENTIONS:
Biological: eOD-GT8 60mer mRNA Vaccine (100µg) — * 2 doses eOD-GT8 60mer mRNA Vaccine (100µg), 2 vaccinations, 8 weeks apart
  * No control group. There is no blinding and no randomization in this open label study

SUMMARY:
A Phase 1 Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) in HIV-1 Uninfected Adults in Good General Health.

DETAILED DESCRIPTION:
A Phase 1 Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) in HIV-1 Uninfected Adults in Good General Health. The hypothesis is that eOD-GT8 60mer mRNA Vaccine as a "germline-targeting" immunogen will generate detectable VRC01-class IgG B-cells in African populations. Eighteen participants. An over-enrollment of up to 2 participants will be permitted to facilitate rapid enrollment. Participants who leave the study for any reason will not be replaced. Adults ≥18 and ≤50 years of age who meet all protocol inclusion criteria, who do not meet any protocol exclusion criteria, who understand the study (as demonstrated by the Assessment of [Informed Consent] Understanding [AOU]), and who can provide written informed consent. Administration of eOD-GT8 60mer mRNA Vaccine (100µg) will occur on Week 0 and Week 8. There is no blinding and no randomization in this open-label study. Participants will be screened up to 56 days before the first IP administration and will be actively followed for 6 months after the last IP administration.

The total study duration including screening and enrollment is approximately 13 months. A participant is expected to be in the study for 10 months from screening to last study visit. The study is expected to screen and enroll over 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults as assessed by a medical history, physical examination, and laboratory tests who are at least 18 years at the time of screening and less than 51 years at the time of first IP administration;
2. Willing to comply with the requirements of the protocol and be available for follow-up for the planned duration of the study;
3. In the opinion of the PI or designee and based on Assessment of (informed consent) Understanding (AOU) results, has understood the information provided and potential impact and/or risks linked to IP administration and participation in the study; written informed consent will be obtained from the participant before any study-related procedures are performed;
4. Willing to undergo HIV testing, risk reduction counselling and receive HIV test results;
5. All women of reproductive potential who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception at least 4 weeks prior to the first IP administration and for 4 months following the last IP administration. Effective contraception includes:

   * Intrauterine device
   * Hormonal contraception, including contraceptive implant or injectable
   * Successful vasectomy in the male partner (considered successful if a woman reports that a male partner has documentation of azoospermia by microscopy [1 year ago], or a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy)
   * Not of reproductive potential, such as having undergone hysterectomy, bilateral oophorectomy or tubal ligation, postmenopausal (≥45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/L), surgically sterile Note: More restrictive measures may be required by the study sites.
6. All participants born female who are not heterosexually active at screening must agree to utilize an effective method of contraception if they become heterosexually active as outlined above;
7. All participants born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Activities (SOAs) (APPENDIX A or APPENDIX B);
8. All sexually active participants born male, regardless of reproductive potential, must be willing to use an effective method of contraception (such as consistent condom use) from the day of the first IP administration until at least 4 months after the last IP administration; Note: For Center for Family Health Research (CFHR) site, males in monogamous relationships whose partners are on a documented and effective contraceptive method will be exempt from this requirement.
9. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to IP-induced antibodies, until the anti-HIV antibody titers become undetectable.

Exclusion Criteria:

1. Positive test for HIV-1 or HIV-2 infection;
2. Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, antituberculosis or other medications considered significant by the Investigator within the previous 6 months; Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single IP administration) of corticosteroid for a non-chronic condition (based on Investigator clinical judgment) at least 2 weeks prior to enrolment in this study.
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the Investigator makes the participant unsuitable for participation in the study;
4. History of substance abuse or alcohol abuse;
5. Reported behaviour that puts the participant at risk for HIV infection within 6 months prior to screening, as defined by:

   * Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection or a casual partner (i.e., no continuing established relationship)
   * Engaged in sex work
   * Frequent excessive daily alcohol use or frequent binge drinking, or any other use of illicit drugs
   * History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus-2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B-or hepatitis C;
   * Two or more sexual partners
6. If female, pregnant or planning a pregnancy during the period of enrolment until 4 months after the last IP administration; or lactating;
7. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions) Note: A participant who states that he or she has easy bruising or bleeding but does not have a formal diagnosis and has IM vaccinations and blood draws without any adverse experience is eligible;
8. Infectious disease diagnosis: chronic hepatitis B-infection (HBsAg-positive), hepatitis C infection (HCV Ab-positive), or active syphilis (screening and confirmatory tests);
9. History of splenectomy;
10. Any of the following abnormal laboratory parameters listed below at screening:

    Hematology
    * Hemoglobin <12.0 g/dl or <7.5 mmol/L
    * Absolute Neutrophil Count (ANC) - ≤1,000/mm3 or < 1.0 x 109 cells/L
    * Absolute Lymphocyte Count (ALC) - ≤650/mm3 or < 0.65 x 109 cells/L
    * Platelets - <125,000 cells/mm3 or <125 x 109 cells/L Chemistry
    * Creatinine - >1.1 x upper limit of normal (ULN)
    * AST - >1.25 x ULN
    * ALT - >1.25 x ULN Urinalysis

    Clinically significant abnormal dipstick confirmed by microscopy:

    • Protein = 1+ or more Blood = 2+ or more (not due to menses) and >10 RBCs per high power field When available, the screening laboratory tests will be reviewed by the study physician. Screening laboratory test(s) may be repeated once at the discretion of the PI or designee to investigate any isolated abnormalities. If Urinalysis is the only exclusion criteria that is met, consider repeat urinalysis to confirm.
11. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after IP administration (Exception is live attenuated influenza vaccine which can be given within 14 days); or receipt of other vaccine (including all COVID-19 vaccinations) within the previous 14 days or planned receipt within 14 days after IP administration; Note: COVID-19 vaccinations: Participants should not have received any COVID-19 vaccinations in the 14 days before or 14 days after IP administration.
12. Receipt of blood transfusion or blood-derived products within the previous 3 months;
13. Participation in another clinical study of an IP currently, within the previous 3 months or expected participation during this study; concurrent participation in an observational study not requiring blood or tissue sample collection is not an exclusion; Note: COVID-19 immunoprophylaxis will be permitted prior to and/or during the study provided the agent has received either Emergency Use Approval by FDA, Conditional Marketing Authorization by the European Medicines Agency, or granted licensure by a country's regulatory agency.
14. Prior receipt of any investigational HIV vaccine candidate or HIV monoclonal antibody Note: Receipt of placebo in a previous HIV vaccine study or monoclonal antibody study will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval.
15. History of significant local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration); (This includes individuals with history of anaphylaxis and/or severe hypersensitivity reaction to mRNA vaccines or its excipients)
16. Psychiatric condition that compromises the safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years;
17. Seizure disorder: A participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years);
18. History of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of completely excised malignancy that is considered cured is not an exclusion);
19. Active, serious infections requiring antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment;
20. Body mass index (BMI) ≥35;
21. Body weight <110 pounds (50 kg);
22. Prior daily use of NSAID/aspirin that cannot be held for 5 days prior to the leukapheresis procedure (if applicable at the study site);
23. If, in the opinion of the PI, it is not in the best interest of the participant to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of eOD-GT8 60mer mRNA Vaccine | 16 months
  To evaluate the safety and tolerability of eOD-GT8 60mer mRNA Vaccine, including local and systemic solicited AEs from Day 1 to Day 7 inclusive after each IP administration, Grade 2 or higher unsolicited AEs from the day of each IP administration through 28 days after, participants with SAEs throughout the study period and participants with MAAEs and AESIs from the first day of IP administration through 24 weeks post final IP administration

CONTACTS AND LOCATIONS:
Locations (2):
- Center for Family Health Research, Kigali, Rwanda
- Aurum Tembisa Clinical Research Centre, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
This will be done with the clinical trial team, collaborators and funding agencies. Also, as information becomes available, this will be shared with the site and study participants. Results dissemination plans will be developed and implemented as the study progresses.
Supporting Information: Study Protocol
Time Frame: Information will be shared as soon as results are publicly available for the investigational product being used in similar studies conducted in other regions. The existing results and data upon which the G003 study is based is yet to be made fully publicly available.
Access Criteria: Access to data will be determined by the study team, partners and funding agencies.
URL: http://www.iavi.org/newsresources/press-releases/2021/first-in-human-clinicaltrial-confirms-novel-hivvaccine-approachdeveloped-by-iavi-andscripps-research

REFERENCES:
- [Derived] Libera M, Caputo V, Laterza G, Moudoud L, Soggiu A, Bonizzi L, Diotti RA. The Question of HIV Vaccine: Why Is a Solution Not Yet Available? J Immunol Res. 2024 Apr 8;2024:2147912. doi: 10.1155/2024/2147912. eCollection 2024. PMID 38628675